CLINICAL TRIAL: NCT07114055
Title: Effect of Ebastine in Patients With Diarrhea Predominant Irritable Bowel Syndrome
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Md. Hazrat Ali (Other)
Responsible Party: Sponsor-Investigator, Md. Hazrat Ali, Principal Investigator, Dhaka Medical College
Organization: Dhaka Medical College (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB-DMC/2025/52
Record Dates: First submitted 2025-07-08; First posted 2025-08-11 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Irritable Bowel Syndrome - Diarrhoea
Keywords: Ebastine
MeSH Terms: interventions — ebastine

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ebastine (Active Comparator): Tab. Ebastine 20mg once daily at night
  Interventions: Drug: ebastine
- Placebo (Placebo Comparator): Tab. Placebo once daily at night
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ebastine — Tab. Ebastine 20mg once daily at night
  Arms: Ebastine
Drug: Placebo — Tab. Placebo once daily at night
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to assess and compare the effect of ebastine and placebo in improving symptoms in patients with diarrhea predominant IBS. It will also assess about the safety of drugs ebastine and placebo by recording the patient reported adverse events. The main questions it aim to answer are:

Does drug ebastine and placebo has any effect on patients with IBS-D? What medical problems do participants have when taking drug ebastine and placebo? Researcher will compare effect of drug ebastine and placebo .

Participant will:

Take drug ebastine 20 mg at night and placebo once daily at night every day for 8 weeks along with lifestyle modifications. After that all two groups will visit the hospital 4 weekly, and their symptoms will be assessed by IBS symptom severity score (IBS-SSS) at baseline, week 4 and week 8. Additionally, patient reported adverse events will be documented.

ELIGIBILITY:
Inclusion criteria

* Age 18 and above
* Patients who meet the Rome IV criteria for IBS-D.

Exclusion criteria

* Presence of alarm features: anemia, weight loss, per rectal bleeding, nocturnal frequency, and family history of colonic cancer
* History of major gastrointestinal surgery
* Medical disease that affect the digestive system, such as uncontrolled diabetes, hyperthyroidism, hypothyroidism
* Pregnant and lactating women
* Vehicle drivers, mechanical operators and aerial operators
* Drug abuse or alcohol abuse

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-15 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
1. Improvement of diarrhea predominant IBS symptoms | [At baseline before randomization and then at week 4, and 8 ]
  The improvement of IBS symptoms will be assessed by IBS symptom severity score (IBS-SSS). This score is a Likert scale with seven domains divided into two parts. Part one is the severity score containing four domains, where domain one has two separate scoring scale. Each scale scoring from 0 to 100, that makes it a total score of 500. The severity is denoted as Mild (Score 75 to 175), Moderate (Score 176 to 300), and severe (Score more than 300). The part two is a descriptive questionnaire about bowel habit.

SECONDARY OUTCOMES:
The effect of ebastine in diarrhea predominant IBS patients | [At baseline before randomization and then at week 4, and 8]
  The improvement of IBS symptoms will be assessed by IBS symptom severity score (IBS-SSS). This score is a Likert scale with seven domains divided into two parts. Part one is the severity score containing four domains, where domain one has two separate scoring scale. Each scale scoring from 0 to 100, that makes it a total score of 500. The severity is denoted as Mild (Score 75 to 175), Moderate (Score 176 to 300), and severe (Score more than 300). The part two is a descriptive questionnaire about bowel habit.
The effect of placebo in diarrhea predominant IBS patients | At baseline before randomization and then at week 4, and 8
  The improvement of IBS symptoms will be assessed by IBS symptom severity score (IBS-SSS). This score is a Likert scale with seven domains divided into two parts. Part one is the severity score containing four domains, where domain one has two separate scoring scale. Each scale scoring from 0 to 100, that makes it a total score of 500. The severity is denoted as Mild (Score 75 to 175), Moderate (Score 176 to 300), and severe (Score more than 300). The part two is a descriptive questionnaire about bowel habit.
Compare the effect of ebastine and placebo | At baseline before randomization and then at week 4, and 8
  The improvement of IBS symptoms will be assessed by IBS symptom severity score (IBS-SSS). This score is a Likert scale with seven domains divided into two parts. Part one is the severity score containing four domains, where domain one has two separate scoring scale. Each scale scoring from 0 to 100, that makes it a total score of 500. The severity is denoted as Mild (Score 75 to 175), Moderate (Score 176 to 300), and severe (Score more than 300). The part two is a descriptive questionnaire about bowel habit.
Adverse events | through study completion, an average of 1 year
  Patient reported adverse events will be documented

CONTACTS AND LOCATIONS:
Locations (1):
- Dhaka Medical College, Dhaka, Bangladesh